CLINICAL TRIAL: NCT02754323
Title: Feasibility Study and Validation of Measuring Apparatus Codesna Stress at Work
Acronym: codesna
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-AOI-08; 2015-A00512-47 (Other: ANSM)
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Stress, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apparatus CODESNA (Other): correlation between job stress measurement by the Maslach Burnout INVENTORY and KARASEK questionnaires and measurement of chronic stress by CODESNA tool
  Interventions: Device: Apparatus CODESNA

INTERVENTIONS:
Device: Apparatus CODESNA — The inclusion period is evaluated at one month and the participation of each patient is two days. One day or the subject performs the evaluation of chronic stress by CODESNA and following through questionnaires and another day to 3 weeks / one month apart, to perform a second chronic stress measurement with tool CODESNA to evaluate its reproducibility and reliability.

SUMMARY:
There are different definitions of stress according to each discipline. In psychology, it is defined according to the individual's ability to adapt. The medical approach focuses on the reactions of the body to stress situations. And the organizational approach seeks to define in terms of sources of stress situations. According to a national interprofessional agreement on stress at work in 2008 is defined as a condition that occurs when there is an imbalance between the perception of a person with constraints imposed by its environment and the perception that it has its own resources to cope.

Stress at work

INRS emphasizes prevention to fight against the cost of work stress and seeks to develop methods and tools objectification stressful situations. The social cost of workplace stress would represent 10 to 20% of the expenses of the branch for employment injuries / occupational diseases of the Social Security According to a survey by the European Agency for Safety and Health at Work conducted in 1999, stress is the cause of 50 to 60% of all lost working days. The cost of occupational stress assessed by INRS represent 830 million euros in 2000 in France.

Media coverage of working conditions related suicides has prompted some companies to communicate about work stress and develop actions.

According to the study of Sumer in 2003, 61% of employees have a highly stressful job and 27% complained of work-related health problems.

However, the 2009 survey shows that job stress is a major risk factor for mental health and is associated with decreased job performance. Burnout sets in stages idealistic enthusiasm, stagnation, frustration, apathy. Therefore, it is essential to track the state of chronic stress as soon as possible to prevent burnout.

Stress testing procedures

The major problem is that there is not now comprehensively measure of stress. The measurement models that are available to date, all incomplete, can be classified according to two categories.

First, the general patterns that measure only partially stress but which can be used in any type of fields. One application of self-KARASEK and the imbalance of effort / reward SIEGRIST. These two models are mainly used for epidemiological studies on job stress.

Second, the specific models that provide a more comprehensive measure but we can only use in the area from which they come. These measure specific stressors (organizational, professional and emotional) in the study population.

The main objective of this study is evaluate the feasibility and validate the measurement of chronic stress by CODESNA tool. The method is to compare the measured result by the CODESNA tool to measure stress questionnaires collected by the Maslach Burnout INVENTORY and KARASEK. This method explores finely enough constraints and allows a comparison of national data.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent
* Belong to a social security scheme
* Working at the University Hospital of Nice

Exclusion Criteria:

* occurrence of an event particularly disturbing staff during the last six months
* raises annual leave of more than seven days in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
the measured result by the CODESNA tool | 1 month
  The result of chronic Stress is expressed in% above the value 100. It measures the chronic stress in a universal scale for all human beings and using as reference the balance point of the autonomic nervous system.
  This shall be measured from the recording of R-R intervals of an ECG, also called Heart Rate Variability (HRV),,. Then the CODESNA algorithms perform mathematical processing being based physiological principle to deliver information Chronic Stress
the measured stress questionnaires collected by the Maslach Burnout INVENTORY scale | 1 Month
  The result of the Maslach Burnout INVENTORY scale is a score
the measured stress questionnaires collected by the KARASEK scale | 1 month
  The result of the KARASEK scale is a score